CLINICAL TRIAL: NCT06068985
Title: Classifying for HER2 Dependence to De-Escalate Neoadjuvant Chemotherapy in Patients With HER2+ Early Breast Cancer Undergoing HER2 Double-Blockade
Acronym: CHERRY-PICK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Roche Pharma AG (Industry); Oncoclínicas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0721; ML44079 (Other Grant/Funding Number: Roche Pharma AG)
Record Dates: First submitted 2023-09-19; First posted 2023-10-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PHESGO™-Based Neoadjuvant Therapy for HER2-Positive Early Breast Cancer (Experimental): This is a single-arm phase II neoadjuvant study using PHESGO™. Participants will receive three cycles of neoadjuvant PHESGO™, with a specific dosage regimen. After three cycles, participants will be reevaluated based on their PET-CT response. PET-CT response is defined as a ≥40% reduction in SUVMax without metabolic progression in non-target lesions. Responders will receive 5 additional cycles of PHESGO™ before surgery. Non-responders will exit the study, following institutional guidelines. Local surgery follows 8 cycles. Adjuvant therapy varies based on pCR status: 1 year of PHESGO™ for pCR; T-DM1 for 14 cycles or investigator's choice chemotherapy plus 10 additional adjuvant cycles of PHESGO™ for non-pCR cases.
  Interventions: Drug: PHESGO

INTERVENTIONS:
Drug: PHESGO — Subcutaneous formulation with pertuzumab and trastuzumab.

SUMMARY:
This study aims to identify HER2-positive early-stage breast cancer patients who could benefit from neoadjuvant treatment using PHESGO™ (pertuzumab and trastuzumab) without chemotherapy. The approach involves utilizing specific biomarkers (HR and HER2 IHC status) to select participants whose tumors strongly rely on the HER2 pathway, potentially benefiting from a HER2-targeted approach without chemotherapy concurrently.

DETAILED DESCRIPTION:
This is a nonrandomized phase II single arm study to assess de-escalation of chemotherapy in participants with HER2-positive early breast cancer undergoing neoadjuvant therapy with PHESGO™. Participants will be evaluated by central laboratory review for confirmation of selected biomarkers (pre-screening). Participants who meet the biomarker assessment criteria will follow the eligibility criteria assessment. Participants with HER2 positive disease that meet the eligibility criteria will be treated with neoadjuvant PHESGO™.

A baseline PET/CT will be performed prior to start of PHESGO™ treatment. All participants will receive fixed-dose subcutaneous formulation with pertuzumab and trastuzumab (PHESGO™) every 21 days for 3 cycles to evaluate PET/CT response. After the 3rd cycle, participants achieving PET/CT response (defined in this trial as ≥40% reduction in the SUVMax as calculated by the formula SUVbaseline SUVresponse/SUVbaseline) will continue treatment with PHESGO™ for 5 additional cycles, completing 8 neoadjuvant cycles of PHESGO™. Participants without PET/CT response after 3rd cycle will be out of study and will receive treatment and surgery according to institutional standard of care. For this cohort of participant, data regarding treatment received, pCR status and outcomes will be collected.

Definitive breast cancer surgery will be performed after the 8th cycle of therapy. After surgery, participants will receive adjuvant treatment according to their response. Participants achieving pCR will receive PHESGO™ alone as adjuvant treatment to complete a total of one year of therapy, thus receiving 10 cycles of adjuvant PHESGO™. Participants not achieving pCR will receive one of two adjuvant therapy options as per investigator's choice: (1) 14 cycles of trastuzumab emtansine (T-DM1), or (2) investigator's choice chemotherapy regimen (up to 6 cycles) plus 10 cycles of PHESGO™. Disease status and survival data collection will be abstracted from medical records for up to 5 years after surgery.

Participants will be followed for recurrence and survival data with abstraction of data from medical records every 3 months in first year after surgery; every 4 months in second and third years; and then annually until five years. Medical procedures and therapies in the follow-up period are not a formal investigational part of this clinical trial and therefore will be performed according to the institutional standard of care.

ELIGIBILITY:
Prescreening Eligibility Criteria (Molecular Assessment):

* Signed prescreening informed consent form (ICF); Women between 18-80 years of age at time of signing ICF.
* ECOG ≤ 1.
* HER2+ breast cancer with clinical stage at presentation: T1cN1, T2, N0-1
* HER2 3+ by IHC
* ER IHC ≤10%
* PR IHC negative (<1%)
* Patients must NOT have received any previous systemic therapy for treatment or prevention of breast cancer.
* Must be willing to provide a tumor tissue sample (archival or recently collected).
* Patients undergoing molecular prescreening will be centrally reviewed for HER2 and hormone receptor status by IHC. These results will be used to verify eligibility in the interventional part of this study.

Inclusion Criteria:

* Signed ICF; Women between 18-80 years of age at time of signing ICF.
* ECOG ≤ 1
* HER2+ breast cancer with clinical stage at presentation: T1cN1, T2, N0-1
* HER2 3+ by IHC, with strongly positive staining for HER2 protein in ≥ 80% of cells, and absence of HER2 negative areas in the tumor
* ER IHC ≤10%
* PR IHC negative (<1%) or 0% of tumor cell nuclei
* Tumors must have at least 10mm measured by breast echography and be assessable for SUVMax (maximum standardized uptake value (SUVmax) ≥ 2.5) using 18FDG-PET-CT scan on baseline imaging.
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue block for central confirmation of HER2 and hormone receptor status and additional biomarker research.
* Baseline LVEF ≥ 55% measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA).
* For women of childbearing potential (WOCBP) who are sexually active: agreement to remain abstinent (refrain from heterosexual intercourse) or use one highly effective non-hormonal contraceptive method with a failure rate of < 1% per year, or two effective non-hormonal contraceptive methods during the treatment period and for 7 months after the last dose of HER2-targeted therapy, and agreement to refrain from donating eggs during this same period.
* A negative serum pregnancy test must be available prior to randomization for WOCBP (premenopausal women and women < 12 months after the onset of menopause), unless they have undergone surgical sterilization (removal of ovaries and/or uterus)

Exclusion Criteria:

* Patients with metastatic disease.
* Any previous systemic chemotherapy or anti-HER2 targeted therapy directed to breast cancer.
* Patients with clinical N2 or N3 disease, T4, or inflammatory breast cancer.
* Concurrent serious diseases that may interfere with planned treatment.
* Patients with a history of concurrent or previously treated non-breast malignancies except for appropriately treated 1) non-melanoma skin cancer and/or 2) in situ carcinomas, including cervix, colon, and skin. A patient with previous invasive non-breast cancer is eligible provided he/she has been disease free for more than 5 years.
* Patients who have received any previous systemic therapy (including chemotherapy, immunotherapy, HER2-targeted agents, endocrine therapy (selective estrogen receptor modulators, aromatase inhibitors, and antitumor vaccines) for treatment or prevention of breast cancer.
* Patients who have a history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) if they have received any systemic therapy for its treatment, or radiation therapy to the ipsilateral breast. Patients are allowed to enter the study if treated with surgery alone.
* Patients with high-risk for breast cancer who have received chemopreventive drugs in the past are not allowed to enter the study.
* Patients with bilateral breast cancer.
* Patients who have undergone an excisional biopsy of primary tumor and/or axillary lymph nodes.
* Axillary lymph node dissection (ALND) or Sentinel lymph node biopsy (SLNB) prior to initiation of neoadjuvant therapy. Patients with clinically negative axilla (by physical examination and radiographic imaging) may undergo a core or needle biopsy procedure prior to neoadjuvant systemic therapy.
* Treatment with any investigational drug within 28 days prior to randomization.
* Serious cardiac illness or medical conditions.
* Inadequate bone marrow function.
* Impaired liver function.
* Inadequate renal function.
* Current severe, uncontrolled systemic disease that may interfere with planned treatment (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease; wound-healing disorders).
* Any major surgical procedure unrelated to breast cancer within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment.
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 7 months after the last dose of HER2-targeted therapy. Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study drug.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study.
* Known active liver disease, for example, active viral hepatitis infection (i.e., hepatitis B or hepatitis C), autoimmune hepatic disorders, or sclerosing cholangitis.
* Concurrent, serious, uncontrolled infections, or known infection with HIV.
* Known hypersensitivity to study drugs, excipients, and/or murine proteins.
* Current chronic daily treatment with corticosteroids (dose > 10 mg methylprednisolone or equivalent excluding inhaled steroids).
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, colon, skin, and/or non-melanoma skin carcinoma.
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe LVSD, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | After eight neoadjuvant cycles of PHESGO™ (each cycle is 21 days)
  This outcome measures the rate of participants with HER2-positive early breast cancer who achieve a pathologic complete response (pCR) following neoadjuvant treatment with PHESGO™ without concurrent chemotherapy. Participants selected based on high HER2 pathway dependence and demonstrating a favorable PET-CT response after the third therapy cycle are evaluated for the absence of residual invasive tumor cells in the breast and lymph nodes.

SECONDARY OUTCOMES:
Rate of Favorable PET-CT Response | After three neoadjuvant PHESGO™ cycles (each cycle is 21 days)
  Measures the percentage of participants showing a ≥40% reduction in SUVMax on PET-CT after three cycles of neoadjuvant PHESGO™. Responders demonstrate significant SUVmax reduction with no metabolic progression in non-target lesions.
Pathologic Response via Residual Cancer Burden (RCB) | Immediately after the end of treatment
  Evaluates pathologic response using the Residual Cancer Burden (RCB) tool, available at the provided link. RCB is assessed to determine the extent of residual cancer after treatment, aiding in treatment response evaluation.
Objective Response Rate by PERCIST 1.0 | After three neoadjuvant PHESGO™ cycles (each cycle is 21 days)
  Measures the percentage of participants achieving complete metabolic response (CMR) or partial metabolic response (PMR) as per PERCIST 1.0 criteria, assessed by site radiology review after three cycles of neoadjuvant PHESGO™. Metabolic response assessment follows the Radiology Assessment section guidelines.
Objective Response Rate by RECIST 1.1 | After eight neoadjuvant cycles of PHESGO™ (each cycle is 21 days)
  Measures the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria from enrollment to eight cycles of neoadjuvant PHESGO™, among those who complete neoadjuvant treatment. Evaluation will be conducted by the local investigator in accordance with RECIST criteria version 1.1.
Invasive Disease-Free Survival (iDFS) Stratified by pCR | From enrollment until an event related to invasive disease occurs, stratified by pCR, assessed up to 5 years
  Measures the time from enrollment to any occurrence of invasive disease, stratified by the presence or absence of pathologic complete response (pCR). Events for iDFS include death from any cause, locoregional or distant recurrence, new breast cancer (ipsilateral or contralateral), and second primary invasive cancer. Invasive breast cancer ipsilateral to the treatment disease is considered a recurrence. Data will be recorded regardless of therapy withdrawal after the first dose. Participants without these events at analysis times will be censored at the latest assessment date.
Event-Free Survival (EFS) Stratified by pCR | From enrollment until an event related to EFS occurs, stratified by pCR, assessed up to 5 years
  Measures the time from enrollment to the occurrence of specific events, stratified by the presence or absence of pathologic complete response (pCR). Events for EFS include death from any cause, locoregional or distant recurrence, new breast cancer (ipsilateral or contralateral), cancer progression, and second primary invasive cancer. Invasive breast cancer ipsilateral to the treatment disease is considered a recurrence. Data will be recorded regardless of therapy withdrawal after the first dose. Participants without these events at analysis times will be censored at the latest assessment date.
Overall Survival (OS) Stratified by pCR | From enrollment until the participant's demise from any cause, assessed up to 5 years
  Measures the time from enrollment to death due to any cause among PET responder participants, stratified by the presence or absence of pathologic complete response (pCR). Participants who have not passed away at the time of analysis will be censored based on the last recorded date when they were known to be alive. Causes of death will be recorded for comprehensive analysis.
Cardiac Events and Left Ventricular Systolic Dysfunction | Through study completion, an average of 5 years
  Evaluates cardiac events in participants, including symptomatic ejection fraction decrease leading to heart failure (NYHA Class III or IV) with a drop in LVEF of at least 10-percentage points from baseline and below 50%. It also assesses cardiac death rates, distinguishing between definite and probable cardiac deaths. Additionally, it monitors the incidence of asymptomatic or mildly symptomatic left ventricular systolic dysfunction (NYHA Class II), defined by a significant LVEF decrease confirmed by a second assessment within approximately 3 weeks.
Safety - Adverse Events | Through study completion, an average of 5 years
  Monitors clinical and laboratory adverse events (AEs) in participants according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Summarizes AEs and includes previously known adverse events related to the medications in the study, categorized as Adverse Events of Special Interest (AESI) per the defined Adverse Events Definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Simon, Principal Investigator — Oncoclínicas
Locations (14):
- Brazil (14):
  - Núcleo de Oncologia da Bahia - NOB (Oncoclínicas), Salvador, Estado de Bahia
  - Centro de Câncer de Brasília - CETTRO (Oncoclínicas), Brasília, Federal District
  - Oncocentro Belo Horizonte (Oncoclínicas), Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Vencer & Oncoclínica, Teresina, Piauí
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital da Fundação Oswaldo Aranha - HFOA, Volta Redonda, Rio de Janeiro
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS - CPO, Porto Alegre, Rio Grande do Sul
  - Universidade Estadual de Campinas - UNICAMP, Campinas, São Paulo
  - Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, São Paulo
  - Centro de Pesquisa do Hospital Pérola Byington, São Paulo, São Paulo
  - A.C. Camargo Cancer Center, São Paulo, São Paulo
  - Centro Paulista de Oncologia (Oncoclínicas), São Paulo, São Paulo
  - Hospital de Amor de Barretos, São Paulo, São Paulo